CLINICAL TRIAL: NCT05832619
Title: Intradermal Acupuncture Versus Sham Acupuncture and SSRI for Treating Adolescents With Major Depressive Disorder: a Study Protocol for a Randomized Controlled Trial
Brief Title: Intradermal Acupuncture Versus Sham Acupuncture and SSRI for Treating Adolescents With Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaomei Shao (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZX010-YA
Record Dates: First submitted 2023-04-15; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Intradermal Acupuncture; Randomized Controlled Trial; Adolescent
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waiting list group (Other): This group will include 40 patients with MDD who will be treated with oral SSRIs only, the dosage of which will be determined by the psychiatrist. After 6 weeks, patients could choose 6 weeks' intradermal acupuncture treatments free of charge.
  Interventions: Drug: SSRI
- SIA+SSRIs group (Sham Comparator): This group will include 40 patients with MDD who will be treated with sham intradermal acupuncture combined with SSRIs. Acupoints related to MDD will be stimulated by acupuncturists and the dosage of oral SSRIs will be determined by the psychiatrist.
  Interventions: Drug: SSRI; Device: SIA
- AIA+SSRIs group (Experimental): This group will include 40 patients with MDD who will be treated with active intradermal acupuncture combined with SSRIs. Acupoints related to MDD will be stimulated by acupuncturists and the dosage of oral SSRIs will be determined by the psychiatrist.
  Interventions: Drug: SSRI; Device: AIA

INTERVENTIONS:
Drug: SSRI — SSRIs antidepressants, including fluoxetine, paroxetine, sertraline, citalopram, etc., will be administered at oral doses determined by the psychiatrist. Once daily for 6 weeks.
  Other Names: selective 5-hydroxytryptamine reuptake inhibitors
Device: SIA — This study will select 4 acupoints (all taken bilaterally) commonly used to treat MDD, namely Taichong (LR3), Neiguan (PC6), Sanyinjiao (SP6) and Shenmen (HT7). The SIA will use the same size, colour and material as the AIA with a thin silicone pad in the middle instead of the needle body. SIA will be attached to the acupoints and retained for 72 hours, removed and rested for one day. A total of 10 sessions will be performed over a period of 6 weeks.
  Other Names: sham intradermal acupuncture
  Arms: SIA+SSRIs group
Device: AIA — This study will select 4 acupoints (all taken bilaterally) commonly used to treat MDD, namely Taichong (LR3), Neiguan (PC6), Sanyinjiao (SP6) and Shenmen (HT7). Depending on acupoints' location, a φ0.20*1.5mm or φ0.20*1.2mm AIA will be selected. Press the AIA to insert it vertically into the acupoint and retain it in the skin. AIA will be retained for 72 hours with a day's rest after removal. During the period of needle retention, participants will be instructed to press the AIA 3-4 times a day for approximately 1 minute each time, with as much stimulation as the patient can tolerate, at intervals of approximately 4 hours. A total of 10 sessions will be performed over a period of 6 weeks.
  Other Names: active intradermal acupuncture
  Arms: AIA+SSRIs group

SUMMARY:
Major depressive disorder (MDD) is a prevalent mental illness characterised by influencing the health and quality of life of patients，often manifesting in individuals under the age of 18. It has been wildly confirmed that acupuncture alone or in combination with the applicable adjuvant therapy for MDD can not only relieve patients' physical symptoms, but also enhance sleep quality. Intradermal acupuncture, as an acceptable and long-lasting treatment modality, is the focus of this research. This study was conducted to investigate the efficacy of intradermal acupuncture in the treatment of MDD.

DETAILED DESCRIPTION:
This study will enroll a total of 120 adolescents with MDD who meet the inclusion criteria. Participants will be randomly assigned 1:1:1 to the waiting list group (patients in this group will be treated with selective 5-hydroxytryptamine reuptake inhibitors (SSRIs) only), sham intradermal acupuncture combined with SSRIs (SIA) group and active intradermal acupuncture combined with SSRIs (AIA) group. The study is aim to evaluate the efficacy of intradermal acupuncture for MDD and examine whether intradermal acupuncture reduces side effects and improves the efficacy of SSRIs for MDD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MDD according to the International Classification of Disease-10 (ICD-10); HAMD-17≥7
2. Aged between 12 and 17 years (no limitation on gender);
3. Take SSRI for at least two weeks;
4. Written informed consent is obtained by the person or guardian.

Exclusion Criteria:

1. ICD-10 diagnoses: schizophrenia, bipolar disorder, manic episode or other psychotic disorders; alcohol and drug addiction;
2. Significant skin lesions, severe allergic diseases, tumors, and severe or unstable internal diseases involving the cardiovascular, digestive, endocrine, or hematological system;
3. Acute suicidal tendency;
4. Allergy to adhesive tape and fear of intradermal acupuncture;
5. Pregnancy and lactation;
6. Mental retardation and difficult to cooperate with doctors.
7. Participating in other clinical trials.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Hamilton Depression Scale-17 (HAMD-17) Scores | [Time Frame: Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.]
  The HAMD scale is the most commonly used in the clinical assessment of depression, including 17 items. The higher the score, the more severe the depression. 0-7 means no depressive symptoms, 8-17 means mild depression, 18-24 was divided into moderate depression, and 25-52 was divided into severe depression.

SECONDARY OUTCOMES:
Changes in the Self-Rating Depression Scale (SDS) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up
  The standard score is the total of all scores multiplied by 1.25 to the nearest whole number on this scale, which has 20 questions. A standard score below 50 is normal; 50-60 is mild depression; 61-70 is moderate depression; 70 or more is severe depression.
Changes in the Pittsburgh Sleep Quality Index (PSQI) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up
  The PSQI is used to assess the sleep quality of the participant in the last 1 month and consisted of 19 self-rated and 5 other rated items. The higher the score, the worse the sleep quality. Sleep quality is divided into 4 levels according to the total score.
Changes in the Patient Health Questionaire-9 (PHQ-9) | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up
  The PHQ-9 was used to screen survey respondents for depression. The scale was developed according to the criteria for diagnosing depression in the American Diagnostic and Statistical Manual of Mental Disorders (4th edition) and is a concise, validated self-assessment and screening tool for depression. There are 9 questions, each with a score of 0-3 (none: 0; a few days: 1; more than half the time: 2; almost every day: 3), for a total score of 0-27.
Changes in the Short Form 36 Questionnaire（SF-36） | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up
  The SF-36 scale has been developed by the American Medical Research Group as a universal scale for measuring quality of life and is widely recognized and used internationally. This scale has 8 dimensions to evaluate health-related quality of life, which are divided into two major categories: physical function (PF), physical function (RP), somatic pain (BP), general health (GH), energy (VT), social function (SF), emotional function (RE), and mental health (MH). the SF-36 scale is to a certain extent a better response to patients' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Chen N, Wu X, Tu M, Xiong S, Jin J, Qu S, Pei S, Fang J, Shao X. Optimizing Treatment for Major Depressive Disorder in Adolescents: The Impact of Intradermal Acupuncture - A Randomized Controlled Trial Protocol. Neuropsychiatr Dis Treat. 2023 Aug 23;19:1819-1832. doi: 10.2147/NDT.S420489. eCollection 2023. PMID 37641586